CLINICAL TRIAL: NCT03216148
Title: A Prospective, Multicentre Trial on the Value of 18F-FET PET in the Post-therapeutic Evaluation of Childhood Brain Tumours
Brief Title: 18F-FET PET in Childhood Brain Tumours
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, PD Dr. Pablo Hernaiz Driever, Principal Investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FET PET 2010; 2008-005786-60 (EudraCT Number)
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Brain Neoplasm
Keywords: FET PET
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: All pediatric patients with brain Tumor receive a FET-PET Investigation in Addition to conventional MRI at the end of the first-line therapy. In case of Progression or Relapse patients may receive a second FET-PET Investigation in Addition to Routine surveillance MRI.
Oversight: Data Monitoring Committee: No

ARMS (1):
- FET-PET (Experimental): All participating patients will receive a FET PET-scan with intravenous O-(2-[18F]Fluoroethyl)-L-Tyrosine parallel to the routine MRI at the end of the first line therapy (restaging) according to the HIT-protocol Second FET PET: In case of suspected tumour recurrence or progression within the follow-up period of 24 (12) months, the participating patient will receive a second FET PET-scan (parallel to an MRI)
  Interventions: Diagnostic Test: FET-PET

INTERVENTIONS:
Diagnostic Test: FET-PET — All participating patients will receive a FET PET-scan parallel to the routine MRI at the end of the first line therapy (restaging) according to the HIT-protocol Second FET PET: In case of suspected tumour recurrence or progression within the follow-up period of 24 (12) months, the participating patient will receive a second FET PET-scan (parallel to an MRI)
  Other Names: O-(2-[18F]Fluoroethyl)-L-Tyrosine

SUMMARY:
FET PET 2010 is a prospective, multicentre trial aiming to evaluate the additional benefit of FET PET in the assessment of remission after first line therapy and during follow-up

DETAILED DESCRIPTION:
2.1 Primary objective The main objective is to evaluate the relative benefit of FET PET in comparison to the MRI in differentiating biologically active tumour tissue from therapy-related changes in paediatric brain tumours after first line therapy (Δ specificityFET PET to specificityMRT) 2.2 Secondary Objectives To assess sensitivity of FET PET in comparison with the sensitivity of MRI (Δ sensitivityFET PET to sensitivityMRT) To assess the positive and negative predictive values (PPV, NPV) of FET PET in comparison with the PPV and NPV of MRI (Δ PPVFET PET to PPVMRT, Δ NPVFET PET to NPVMRT) To evaluate specificity, sensitivity, PPV, and NPV by SUVratio analyses of FET PET data To evaluate the potential of FET PET for non-invasive tumour grading (WHO I/II vs. III/IV) by kinetic studies when histology is available To assess adverse events and toxicity profile

2.3 Endpoints (Standard of truth1) 2.3.1 Primary Endpoint The primary endpoint is an event free survival of the follow-up period of 24 (12) months after first line therapy (confirmed by clinical and neuroradiological assessment) or the confirmed diagnosis of progression or recurrence of brain tumour tissue (confirmed by histology or clinical and neuroradiological assessment).

The follow-up period for patients with a low risk of tumour recurrence after first line therapy, i.e. astrocytoma WHO grade I-II, oligodendroglioma WHO grade I-II, germ cell tumour, choroid plexus tumour, craniopharyngioma will be 24 months.

The follow-up period for patients with a high risk of tumour recurrence after first line therapy, i.e. astrocytoma WHO grade III-IV, oligodendroglioma WHO grade III-IV, medulloblastoma, supratentorial PNET, AT/RT and other high-grade tumour lesions will be 12 months.

2.3.2 Secondary Endpoints To assess the secondary objectives of the FET PET 2010 study, the investigators will determine event free survival of the follow-up period of 24 (12) months after first line therapy (confirmed by clinical and neuroradiological assessment) or the confirmed diagnosis of progression or recurrence of brain tumour tissue (confirmed by histology or clinical and neuroradiological assessment).

Histopathological characteristics of recurrent tumours (WHO grade I-IV) Safety and Toxicity (evolution according to CTCEA v3.0 criteria): the NCI Common Terminology Criteria for Adverse Events v3.0 is a descriptive terminology, that is used for Adverse Event (AE) reporting. A grading scale is provided for each AE term. Attached is a selection of categories, which are required to assess safety and toxicity of FET PET examinations.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (given by the parents as legal representatives of the patients and given by the patients)
* Completion of the first line therapy according to the current HIT-protocols (Current and subsequent paediatric primary brain tumour treatment studies approved by GPOH)
* Fully evaluable MRI at the end of first line therapy as confirmed by the reference centre of neuroradiology (Prof. Dr. M. Warmuth-Metz, Würzburg)
* Histology of primary brain tumour confirmed by local and reference centre of Neuropathology (Prof. Dr. T. Pietsch) except for patients where tumour diagnosis is confirmed by the reference centre of neuroradiology, i.e. NF-1 and confirmed LGG or patient with diffuse intrinsic pontine glioma
* Laboratory requirements prior to enrolment: Serum creatinine: within normal limits; AST, ALT: not more than 10 x above normal limits
* Age at inclusion: 1 year to 17 years
* Children below the age of 12 years are included as 2 of 3 paediatric patients with a brain tumour are younger than 12 years. Furthermore, young age is a known negative risk factor for different histological entities. Thus, this group is the most likely to benefit from the results of this study
* In all patients with reproductive potential, a pregnancy must be excluded by a pregnancy test before FET PET investigation
* Highly effective contraception in women with reproductive potential (defined as pearl index < 1) during study participation and follow up time
* No participation in other clinical trials according to AMG with the same clinical indication over the course of the FET PET 2010 study

Exclusion Criteria:

* Presence of solid non-CNS tumours or leukaemia
* MRI at completion of first line therapy that does not meet standard quality criteria for evaluation as defined by the reference centre for neuroradiology of the HITNetzwerk (Würzburg, Prof. Warmuth-Metz);
* Known allergic reactions or drug intolerance to contrast agents
* Patients according to § 88 StrhlSchV
* Pregnancy or breast-feeding
* Women (adolescents) of childbearing potential without highly effective contraception (PEARL-Index < 1%), for example ParaGard IntraUterineDevice (IUD), Mirena IUD, Implants, Depo Provera Injections;
* Persons who are detained officially or legally to an official institute

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Differentiating biologically active Tumor tissue from therapy related changes by using MRI (Magnetic Resonance Imaging) and FET PET | 3 years
  The main objective is to evaluate the relative benefit of FET PET in comparison to the MRI in differentiating residual biologically active tumour tissue from therapy related changes in paediatric brain tumours after first line therapy (Δ specificityFET PET to specificityMRT)

SECONDARY OUTCOMES:
Sensitivity of FET-PET when differentiating biologically active Tumor tissue from therapy-related changes by using MRI (Magnetic Resonance Imaging) and FET PET | 3 years
  To assess sensitivity of FET PET in comparison with the sensitivity of MRI (Δ sensitivityFET PET to sensitivityMRT)
Assessment of the predictive value of FET-PET when differentiating biologically active Tumor tissue from therapy-related changes by using MRI (Magnetic Resonance Imaging) and FET PET | 4 years
  (PPV, NPV) of FET PET in comparison with the PPV and NPV of MRI (Δ NPVFET PET to NPVMRT)
Assessment of Tumor grading by FET-PET when differentiating biologically active Tumor tissue from therapy-related changes by using MRI (Magnetic Resonance Imaging) and FET PET | 4 years
  SUVratio analyses of FET PET data to allow for Analysis of Tumor grading when histological results are available
Safety data on FET-PET in children with brain tumors | 3 years
  To assess adverse events and toxicity Profile using Common Terminology Criteria for Adverse Events, CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Hernáiz Driever, MD, Principal Investigator — Charite University, Berlin, Germany; Michail Plotkin, MD, Study Chair — Vivantes Klinikum
Locations (22):
- Germany (22):
  - Klinikum Augsburg, Onkologie, Augsburg
  - Charité Universitätsmedizin Berlin, CVK, Onkologie, Berlin
  - Evangelisches Krankenhaus Bielefeld gGmbH, Onkologie, Bielefeld
  - Universitätsklinikum Bonn, Onkologie, Bonn
  - Klinikum Bremen-Mitte gGmbH, Onkologie, Bremen
  - Uniklinik Köln, Pädiatrische Onkologie, Cologne
  - Kliniken der Stadt Köln gGmbH, Cologne
  - Universitätsklinikum Düsseldorf, Onkologie, Düsseldorf
  - Universitätsklinikum Essen, Onkologie, Essen
  - Klinik für Nuklearmedizin, Freiburg im Breisgau
  - Klinik für Pädiatrische Hämatologie und Onkologie, Freiburg im Breisgau
  - Zentrum für Kinder- und Jugendmedizin, Angelika-Lautenschläger-Klinik, Onkologie, Heidelberg
  - Institut für Neurowissenschaften und Medizin, Physik der medizinischen Bildgebung, Forschungszentrum Jülich, Nuklearmedizin, Jülich
  - Universitätsklinikum Mainz, Onkologie, Mainz
  - Kinderklinik München Schwabing, Onkologie, München
  - Nuklearmedizinische Klinik und Poliklinik, München
  - Klinik für Kinder- und Jugendmedizin - Pädiatrische Hämatologie und Onkologie, Münster
  - Klinik für Nuklearmedizin, Münster
  - Klinikum Stuttgart - Olgahospital, Onkologie, Stuttgart
  - Klinikum Stuttgart, Nuklearmedizin, Stuttgart
  - Universitätsklinikum Tübingen, Onkologie, Tübingen
  - Universitäts-Kinderklinik Würzburg, Würzburg